CLINICAL TRIAL: NCT04986605
Title: The Effectiveness of ECP in Diffuse Cutaneous Systemic Sclerosis
Brief Title: Extracorporeal Photopheresis in Early Diffuse Cutaneous Systemic Sclerosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Principal Investigator, Janet Pope, Head of Rheumatology, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECR-CAN-011068
Record Dates: First submitted 2021-06-01; First posted 2021-08-03 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Diffuse Cutaneous Systemic Sclerosis
Keywords: systemic sclerosis; scleroderma; extracorporeal photopheresis; connective tissue diseases; skin diseases
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Connective Tissue Diseases; Skin Diseases | interventions — Photopheresis; Methoxsalen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Administration of Extracorporeal Photopheresis Treatment (Experimental): Duration of treatment: 48 weeks. Treatments occur on 2 consecutive days every 4 weeks.
  Dose of UVADEX: Treatment Volume x 0.017 = mL of UVADEX for each treatment Treatment Volume (TV) is defined as: The total volume of Buffy Coat plus prime solution that will undergo photoactivation.
  Route of administration: Extracorporeal
  Interventions: Device: Extracorporeal Photopheresis (ECP); Drug: UVADEX

INTERVENTIONS:
Device: Extracorporeal Photopheresis (ECP) — Drug Intervention using a medical device. The ECP device is already licensed in Canada. License No.7703. ECP treatment, using the drug UVADEX, will be given on 2 consecutive days every 4 weeks for a total of 26 treatment days (48 weeks).
  Other Names: ECP; 8-mop
Drug: UVADEX — The phase II aspect of the study refers to the drug, methoxsalen. Methoxsalen is being used off label from the currently approved indications in the monograph. The study is proposing to use methoxsalen in combination with with extracorporeal photopheresis for the treatment of diffuse cutaneous systemic sclerosis. Treatment will be given in addition to standard of care medications for SSc.
  Other Names: 8-mop

SUMMARY:
The purpose of this study is to assess feasibility, safety and preliminary efficacy of Extracorporeal Photopheresis in the treatment of active diffuse cutaneous systemic sclerosis (dcSSc). This pilot study will help to determine if further study (a RCT) is justified.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc, Scleroderma) is a multisystem autoimmune disease characterized by widespread vascular injury and progressive fibrosis of the skin and internal organs. There is no effective treatment for the majority of patients with diffuse scleroderma (diffuse cutaneous systemic sclerosis; dcSSc). Only few therapies have shown modest benefits in regard to some specific organ pathologies. In the early stage of dcSSc, it may be possible to reverse inflammation and reduce the probability of irreversible fibrosis via significant immune modulation as later, often the fibrosis doesn't improve with treatment.

This is a pilot study that will treat 15 participants with dcSSc who meet the eligibility criteria. The objective of the study is to determine if the benefit of Extracorporeal photopheresis (ECP) and safety are favorable in order to consider and help in the design of a randomized controlled trial (RCT). This is a Phase II study that is uncontrolled and patients will remain on their background immunosuppressive treatment unless if contraindicated for safety or drug interactions. The trial is powered to show a mean change in skin thickness measured with modified Rodnan skin score (mRSS) of ≥5 over one year, in an uncontrolled, unblinded study. The Health Assessment Questionnaire Disability Index (HAQ-DI), patient and physician global scores, inflammatory markers, and combined response index in SSc (CRISS) will all be exploratory outcomes. Other outcomes such as changes in cells on skin biopsies from baseline to end of the trial will be explored if the study is positive.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with SSc, aged 18 years or older, and:
2. Subjects must meet the ACR/EULAR classification criteria for SSc (2013).
3. Early dcSSc (within 5 years of first non-Raynaud's phenomenon symptom) or any other dcSSc patients who have at least one of the signs of disease activity: mRSS of 15 or more, presence of tendon friction rubs, elevated inflammatory markers thought to be due to active dcSSc and not related to other issues such as infection or ILD with FVC% predicted <80% or HRCT showing ILD thought to be from SSc.
4. Able to give informed consent.

Exclusion Criteria:

1. Poor pulmonary function (FVC<40% and/or DLCO<30%).
2. Class IV PAH or PH.
3. Clinically significant cardiac disease.
4. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, cardiac, hepatic, pancreatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease; and cancer (i.e. co-existing melanoma, basal cell, or squamous cell skin carcinoma).
5. Chronic or ongoing active infectious disease requiring systemic treatment, including active tuberculosis (TB) infection.
6. Seropositivity for human immunodeficiency virus (HIV) at study entry.
7. Active viral infection with viral replication of hepatitis B or C virus at study entry.
8. Thrombophilia.
9. Contraindications to heparin including history of heparin-induced thrombocytopenia (HIT) or heparin-induced thrombocytopenia and thrombosis (HITTS), history of thrombocytopenia with pentosan polysulfate, known hypersensitivity to heparin or pork products.
10. Low Platelet count (less than 100,000 per mm3).
11. Aphakia (absence or loss of the eye's lens and has not been replaced with an artificial lens), because of the significantly increased risk of retinal damage due to the absence of lenses.
12. Severe anemia (hemoglobin <70g/L).
13. High white blood cell count (greater than 25000 mm3).
14. A history of surgical spleen removal.
15. A history of a light sensitive disease state, i.e. lupus erythematosus, porphyria cutanea tarda, erythropoietic protoporphyria, variegate porphyria, xeroderma pigmentosum and albinism.
16. Previous idiosyncratic reactions to psoralen compounds.
17. Patients who are using photosensitizing drugs such as anthralin, coal tar or coal tar derivatives, griseofulvin, phenothiazines, nalidixic acid, halogenated salicylanilides (bacteriostatic soaps), sulfonamides, tetracyclines, thiazides, and certain organic staining dyes such as methylene blue, toluidine blue, rose bengal and methyl orange.
18. Treatment with more than 2 immunosuppressants (including mofetil mycophenolate, methotrexate, cyclophosphamide, biologics) at study entry.
19. Pregnancy, breast feeding or child bearing potential without practicing highly effective contraception (and partners for men in the study).
20. Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder).
21. Participation in another clinical trial within six weeks before randomization in this study.
22. Previous use of Extracorporeal photopheresis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in skin thickness measured by modified Rodnan Skin Score | 48 weeks
  modified Rodnan Skin Score (mRSS): is a standard outcome measure for skin disease in SSc and calculated by measuring skin thickness in 17 different body sites (each site scored 0-3, with a total possible additive score of 51). A higher skin score (or a higher "skin thickness") and progression of this score, is predictive of internal organ involvement and mortality. While a lower or improving (lessening) score is associated with favorable outcomes, including better survival.

SECONDARY OUTCOMES:
Change in the modified Rodnan Skin Score | 12, 24 and 36 weeks
  modified Rodnan Skin Score (mRSS): is a standard outcome measure for skin disease in SSc and calculated by measuring skin thickness in 17 different body sites (each site scored 0-3, with a total possible additive score of 51). A higher skin score (or a higher "skin thickness") and progression of this score, is predictive of internal organ involvement and mortality. While a lower or improving (lessening) score is associated with favorable outcomes, including better survival.
Combined Response Index in diffuse cutaneous systemic sclerosis score | 24 weeks
  CRISS score: It is calculated according to changes from the start of a study, compared to an endpoint, by using the modified Rodnan Skin Score (mRSS), the Health Assessment Questionnaire - Disability Index (HAQ-DI), patient and physician global assessment of scleroderma-related health, and forced vital capacity. A CRISS score of ≥ 0.6 indicates likelihood that a patient improved on treatment.
  Will be calculated with baseline data and to define disease progression at 6 months.
Change in Forced Vital Capacity | 6 and 12 months
  Change in Pulmonary Function as measured by percentage of Improving or worsening FVC.
  The FVC (Forced vital Capacity) is the total amount of air exhaled during the FEV (Forced expiratory volume) test.
Change in the diffusing capacity for carbon monoxide | 6 and 12 months
  Change in Pulmonary Function as measured by percentage of Improving or worsening DLCO.
  The DLCO (diffusing capacity of the lungs for carbon monoxide) measures the ability of the lungs to transfer gas from inhaled air to the red blood cells in pulmonary capillaries.
Change in physician global assessment of disease activity | 12, 24, 36 and 48 weeks
  Measured on a Visual Analogue Scale (VAS) from 0-10, with 0 being no disease activity and 10 being the worst possible disease activity.
Change in physician global assessment of disease severity | 12, 24, 36 and 48 weeks
  Measured on a Visual Analogue Scale (VAS) from 0-10, with 0 being no disease severity and 10 being the worst possible disease severity.
Change in physician global assessment of disease damage | 12, 24, 36 and 48 weeks
  Measured on a Visual Analogue Scale (VAS) from 0-10, with 0 being no disease damage and 10 being the worst possible disease damage.
Change in patient global assessment of health status | 12, 24, 36 and 48 weeks
  Measured on a Visual Analogue Scale (VAS) from 0-100, with 0 being no overall effect of disease on participant, and 100 being the worst possible overall effect of disease on participant.
  This is a patient reported outcome.
Change in Scleroderma Health Assessment Questionnaire | 12, 24, 36 and 48 weeks
  The SHAQ combines the disability and pain scales of the HAQ (HAQ-DI), with five scleroderma-specific Visual Analogue Scales for: digital ulcers, Raynaud's phenomenon, gastrointestinal (GI) symptoms, lung symptoms, and overall disease severity.
  The HAQ-DI yields a score of 0-3, that indicates the extent of the respondent's functional limitations.
  Each VAS score is scaled from 0 to 3, with 0 being no symptoms and 3 being the worst possible symptom severity.
  A composite VAS score is not created nor are the individual VAS scores incorporated into the HAQ DI score. Typically, each VAS score is reported individually. There is a proposed way to obtain a combined score obtained by pooling the 8 domains of the HAQ DI and the 5 VASs; however, this approach has not yet been widely accepted.
  This is a patient reported outcome.
Change in serum concentrations C-Reactive Protein | 12, 24, 36 and 48 weeks
  Change in serum concentrations of the acute phase reactant, CRP
  CRP aids in the evaluation of stress, trauma, infection, inflammation, surgery & associated diseases. Blood levels of C-Reactive Protein (CRP) are known to rise in acute disease to a level of up to 50 mg/L in the presence of slight to moderate inflammatory process. Values >50 mg/L indicate high and extensive inflammatory activity.
Change in serum concentrations of Erythrocyte Sedimentation Rate | 12, 24, 36 and 48 weeks
  Change in serum concentrations of the acute phase reactant, ESR
  Reference ranges:
  Male: 0-10 mm/h Female: 0-20 mm/h
  A faster-than-normal rate may indicate inflammation in the body. Inflammation is part of the immune response system. The higher the number, the higher the likelihood of inflammation.

OTHER OUTCOMES:
Regimen-related toxicities | assessed for duration of treatment up to 48 weeks, and up to 12 weeks post-treatment
  Adverse Events (AEs) >= Grade 3 and assessed by the investigator as 1 of the following: related or unrelated to treatment
Infectious complications | assessed for duration of treatment up to 48 weeks, and up to 1 month post-treatment
Change in peripheral levels of T-cell activation marker - sIL-2R | 12, 24, 36 and 48 weeks
  interleukin 2 receptor (sIL-2R)
  Serum sIL-2R level is a sensitive and quantitative marker of circulating peripheral blood mononuclear cell activation.
  Normal range of serum sIL-2R is below 2500 pg/ml. High levels may be found in conditions associated with T-cell activation.
Change in peripheral levels of fibrillogenesis - amino terminal propeptide of type III collagen | 12, 24, 36 and 48 weeks
  Amino-terminal propeptide of procollagen type III (PIIINP) is generated during the synthesis of type III collagen. PIIINP is a non-specific marker of soft tissue injury.
  PIIINP in serum has been shown to correlate with fibrillogenesis, and thus to be a potential direct marker of type III collagen deposition.
  PIIINP reference range Adult (>19 years): 1.2 - 4.2 ug/L
Change in CD3-positive cell count (T-cell marker) in skin biopsies of involved forearm skin | 24 and 48 weeks
  Measured by immunohistochemistry (IHC) as the percentage of CD3-positive cells per total number of cells/mm2.
  Reference rage not established (there is no range, we are looking for a stat significant change (decrease) from baseline)
Change in myofibroblast count in skin biopsies of involved forearm skin | 24 and 48 weeks
  Myofibroblasts are cells involved in the inflammatory response to injury. Myofibroblasts play an active role in collagen synthesis, and correlate with clinical measures of disease activity in SSc.
  Measured by immunohistochemistry (IHC) as the percentage of alpha-SMA-positive cells per total number of cells/mm2.
  Reference range not established

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Janet E Pope, MD PhD, Principal Investigator — University of Western Ontario, Division of Rheumatology, St. Joseph's Health Care, London, Ontario, Canada
Locations (1):
- Rheumatology Clinic, St. Joseph's Health Care, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Komocsi A, Vorobcsuk A, Faludi R, Pinter T, Lenkey Z, Kolto G, Czirjak L. The impact of cardiopulmonary manifestations on the mortality of SSc: a systematic review and meta-analysis of observational studies. Rheumatology (Oxford). 2012 Jun;51(6):1027-36. doi: 10.1093/rheumatology/ker357. Epub 2012 Jan 5. PMID 22223705
- [Background] Nihtyanova SI, Schreiber BE, Ong VH, Rosenberg D, Moinzadeh P, Coghlan JG, Wells AU, Denton CP. Prediction of pulmonary complications and long-term survival in systemic sclerosis. Arthritis Rheumatol. 2014 Jun;66(6):1625-35. doi: 10.1002/art.38390. PMID 24591477
- [Background] Young A, Khanna D. Systemic sclerosis: a systematic review on therapeutic management from 2011 to 2014. Curr Opin Rheumatol. 2015 May;27(3):241-8. doi: 10.1097/BOR.0000000000000172. PMID 25775190
- [Background] Kowal-Bielecka O, Veale DJ. DMARDs in systemic sclerosis: do they exist? In: Distler O, ed. Scleroderma-modern aspects of pathogenesis, diagnosis and therapy. Uni-MedVerlag AG: Bremen-London-Boston; 2009: 89-95.
- [Background] Khanna D, Berrocal VJ, Giannini EH, Seibold JR, Merkel PA, Mayes MD, Baron M, Clements PJ, Steen V, Assassi S, Schiopu E, Phillips K, Simms RW, Allanore Y, Denton CP, Distler O, Johnson SR, Matucci-Cerinic M, Pope JE, Proudman SM, Siegel J, Wong WK, Wells AU, Furst DE. The American College of Rheumatology Provisional Composite Response Index for Clinical Trials in Early Diffuse Cutaneous Systemic Sclerosis. Arthritis Rheumatol. 2016 Feb;68(2):299-311. doi: 10.1002/art.39501. PMID 26808827
- [Background] Valentini G, Silman AJ, Veale D. Assessment of disease activity. Clin Exp Rheumatol. 2003;21(3 Suppl 29):S39-41. PMID 12889221
- [Background] Medsger TA Jr, Bombardieri S, Czirjak L, Scorza R, Della Rossa A, Bencivelli W. Assessment of disease severity and prognosis. Clin Exp Rheumatol. 2003;21(3 Suppl 29):S42-6. PMID 12889222
- [Background] Ong VH, Denton CP. Innovative therapies for systemic sclerosis. Curr Opin Rheumatol. 2010 May;22(3):264-72. doi: 10.1097/BOR.0b013e328337c3d6. PMID 20190640
- [Background] Becker MO, Bruckner C, Scherer HU, Wassermann N, Humrich JY, Hanitsch LG, Schneider U, Kawald A, Hanke K, Burmester GR, Riemekasten G. The monoclonal anti-CD25 antibody basiliximab for the treatment of progressive systemic sclerosis: an open-label study. Ann Rheum Dis. 2011 Jul;70(7):1340-1. doi: 10.1136/ard.2010.137935. Epub 2010 Nov 10. No abstract available. PMID 21068100
- [Background] Rook AH, Freundlich B, Jegasothy BV, Perez MI, Barr WG, Jimenez SA, Rietschel RL, Wintroub B, Kahaleh MB, Varga J, et al. Treatment of systemic sclerosis with extracorporeal photochemotherapy. Results of a multicenter trial. Arch Dermatol. 1992 Mar;128(3):337-46. PMID 1550365
- [Background] Knobler RM, French LE, Kim Y, Bisaccia E, Graninger W, Nahavandi H, Strobl FJ, Keystone E, Mehlmauer M, Rook AH, Braverman I; Systemic Sclerosis Study Group. A randomized, double-blind, placebo-controlled trial of photopheresis in systemic sclerosis. J Am Acad Dermatol. 2006 May;54(5):793-9. doi: 10.1016/j.jaad.2005.11.1091. PMID 16635659
- [Background] Enomoto DN, Mekkes JR, Bossuyt PM, Yong SL, Out TA, Hoekzema R, de Rie MA, Schellekens PT, ten Berge IJ, de Borgie CA, Bos JD. Treatment of patients with systemic sclerosis with extracorporeal photochemotherapy (photopheresis). J Am Acad Dermatol. 1999 Dec;41(6):915-22. doi: 10.1016/s0190-9622(99)70246-x. PMID 10570373
- [Background] Oon S, Huq M, Godfrey T, Nikpour M. Systematic review, and meta-analysis of steroid-sparing effect, of biologic agents in randomized, placebo-controlled phase 3 trials for systemic lupus erythematosus. Semin Arthritis Rheum. 2018 Oct;48(2):221-239. doi: 10.1016/j.semarthrit.2018.01.001. Epub 2018 Jan 6. PMID 29426575
- [Background] Pope JE, Baron M, Bellamy N, Campbell J, Carette S, Chalmers I, Dales P, Hanly J, Kaminska EA, Lee P, et al. Variability of skin scores and clinical measurements in scleroderma. J Rheumatol. 1995 Jul;22(7):1271-6. PMID 7562757
- [Background] Clements P, Lachenbruch P, Siebold J, White B, Weiner S, Martin R, Weinstein A, Weisman M, Mayes M, Collier D, et al. Inter and intraobserver variability of total skin thickness score (modified Rodnan TSS) in systemic sclerosis. J Rheumatol. 1995 Jul;22(7):1281-5. PMID 7562759
- [Background] Clements PJ, Lachenbruch PA, Seibold JR, Zee B, Steen VD, Brennan P, Silman AJ, Allegar N, Varga J, Massa M, et al. Skin thickness score in systemic sclerosis: an assessment of interobserver variability in 3 independent studies. J Rheumatol. 1993 Nov;20(11):1892-6. PMID 8308774
- [Background] Furst DE, Khanna D, Mattucci-Cerinic M, Silman AJ, Merkel PA, Foeldvari I; OMERACT 7 Special Interest Group. Scleroderma--developing measures of response. J Rheumatol. 2005 Dec;32(12):2477-80. PMID 16331791
- [Background] Pope JE, Bellamy N. Outcome measurement in scleroderma clinical trials. Semin Arthritis Rheum. 1993 Aug;23(1):22-33. doi: 10.1016/s0049-0172(05)80024-1. PMID 8235663
- [Background] Pope J, McBain D, Petrlich L, Watson S, Vanderhoek L, de Leon F, Seney S, Summers K. Imatinib in active diffuse cutaneous systemic sclerosis: Results of a six-month, randomized, double-blind, placebo-controlled, proof-of-concept pilot study at a single center. Arthritis Rheum. 2011 Nov;63(11):3547-51. doi: 10.1002/art.30549. PMID 21769850
- [Background] Gordon JK, Martyanov V, Franks JM, Bernstein EJ, Szymonifka J, Magro C, Wildman HF, Wood TA, Whitfield ML, Spiera RF. Belimumab for the Treatment of Early Diffuse Systemic Sclerosis: Results of a Randomized, Double-Blind, Placebo-Controlled, Pilot Trial. Arthritis Rheumatol. 2018 Feb;70(2):308-316. doi: 10.1002/art.40358. Epub 2017 Dec 29. PMID 29073351
- [Background] Boyang Z, Nevskaya T, Pope J et al. Improvement in Skin Score after 2 Years in Early Diffuse Cutaneous Systemic Sclerosis (dcSSc) Patients is Associated with Improvement in Multiple Other Domains of Disease Measurement. J Rheumatol 2018 abstract from the Canadian Rheumatology Association February 2020 meeting (Vancouver).
- [Background] Merkel PA, Silliman NP, Clements PJ, Denton CP, Furst DE, Mayes MD, Pope JE, Polisson RP, Streisand JB, Seibold JR; Scleroderma Clinical Trials Consortium. Patterns and predictors of change in outcome measures in clinical trials in scleroderma: an individual patient meta-analysis of 629 subjects with diffuse cutaneous systemic sclerosis. Arthritis Rheum. 2012 Oct;64(10):3420-9. doi: 10.1002/art.34427. PMID 22328195
- [Background] van Laar JM, Farge D, Sont JK, Naraghi K, Marjanovic Z, Larghero J, Schuerwegh AJ, Marijt EW, Vonk MC, Schattenberg AV, Matucci-Cerinic M, Voskuyl AE, van de Loosdrecht AA, Daikeler T, Kotter I, Schmalzing M, Martin T, Lioure B, Weiner SM, Kreuter A, Deligny C, Durand JM, Emery P, Machold KP, Sarrot-Reynauld F, Warnatz K, Adoue DF, Constans J, Tony HP, Del Papa N, Fassas A, Himsel A, Launay D, Lo Monaco A, Philippe P, Quere I, Rich E, Westhovens R, Griffiths B, Saccardi R, van den Hoogen FH, Fibbe WE, Socie G, Gratwohl A, Tyndall A; EBMT/EULAR Scleroderma Study Group. Autologous hematopoietic stem cell transplantation vs intravenous pulse cyclophosphamide in diffuse cutaneous systemic sclerosis: a randomized clinical trial. JAMA. 2014 Jun 25;311(24):2490-8. doi: 10.1001/jama.2014.6368. PMID 25058083
- [Background] Sullivan KM, Goldmuntz EA, Keyes-Elstein L, McSweeney PA, Pinckney A, Welch B, Mayes MD, Nash RA, Crofford LJ, Eggleston B, Castina S, Griffith LM, Goldstein JS, Wallace D, Craciunescu O, Khanna D, Folz RJ, Goldin J, St Clair EW, Seibold JR, Phillips K, Mineishi S, Simms RW, Ballen K, Wener MH, Georges GE, Heimfeld S, Hosing C, Forman S, Kafaja S, Silver RM, Griffing L, Storek J, LeClercq S, Brasington R, Csuka ME, Bredeson C, Keever-Taylor C, Domsic RT, Kahaleh MB, Medsger T, Furst DE; SCOT Study Investigators. Myeloablative Autologous Stem-Cell Transplantation for Severe Scleroderma. N Engl J Med. 2018 Jan 4;378(1):35-47. doi: 10.1056/nejmoa1703327. PMID 29298160
- [Background] Fernandez-Codina A, Walker KM, Pope JE; Scleroderma Algorithm Group. Treatment Algorithms for Systemic Sclerosis According to Experts. Arthritis Rheumatol. 2018 Nov;70(11):1820-1828. doi: 10.1002/art.40560. Epub 2018 Sep 17. PMID 29781586
- [Background] Khanna D, Denton CP, Lin CJF, van Laar JM, Frech TM, Anderson ME, Baron M, Chung L, Fierlbeck G, Lakshminarayanan S, Allanore Y, Pope JE, Riemekasten G, Steen V, Muller-Ladner U, Spotswood H, Burke L, Siegel J, Jahreis A, Furst DE. Safety and efficacy of subcutaneous tocilizumab in systemic sclerosis: results from the open-label period of a phase II randomised controlled trial (faSScinate). Ann Rheum Dis. 2018 Feb;77(2):212-220. doi: 10.1136/annrheumdis-2017-211682. Epub 2017 Oct 24. PMID 29066464
- [Background] Namas R, Tashkin DP, Furst DE, Wilhalme H, Tseng CH, Roth MD, Kafaja S, Volkmann E, Clements PJ, Khanna D; Participants in the Scleroderma Lung Study I and members of the Scleroderma Lung Study II Research Group. Efficacy of Mycophenolate Mofetil and Oral Cyclophosphamide on Skin Thickness: Post Hoc Analyses From Two Randomized Placebo-Controlled Trials. Arthritis Care Res (Hoboken). 2018 Mar;70(3):439-444. doi: 10.1002/acr.23282. Epub 2018 Feb 9. PMID 28544580
- [Background] Gazi H, Pope JE, Clements P, Medsger TA, Martin RW, Merkel PA, Kahaleh B, Wollheim FA, Baron M, Csuka ME, Emery P, Belch JF, Hayat S, Lally EV, Korn JH, Czirjak L, Herrick A, Voskuyl AE, Bruehlmann P, Inanc M, Furst DE, Black C, Ellman MH, Moreland LW, Rothfield NF, Hsu V, Mayes M, McKown KM, Krieg T, Siebold JR. Outcome measurements in scleroderma: results from a delphi exercise. J Rheumatol. 2007 Mar;34(3):501-9. Epub 2007 Feb 1. PMID 17299843
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Csuka ME, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American College of Rheumatology/European League against Rheumatism collaborative initiative. Arthritis Rheum. 2013 Nov;65(11):2737-47. doi: 10.1002/art.38098. Epub 2013 Oct 3. PMID 24122180